CLINICAL TRIAL: NCT05308381
Title: Impact of Different Pre-exercise Breakfast on Post-exercise Glycaemic Response, Appetite and Energy Balance
Brief Title: Breakfast, Exercise and Metabolic Health in Healthy Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Principal Investigator, Yung-Chih Chen, Principal Investigatior, National Taiwan Normal University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 202012HM031-
Record Dates: First submitted 2022-03-16; First posted 2022-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Metabolic Health; Appetitive Behavior; Energy Balance
Keywords: High protein breakfast; postprandial glycaemia; Appetite; Energy balance
MeSH Terms: conditions — Appetitive Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants and Researchers will be blinded to the interventions.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fasted exercise (Experimental): Fasted prior to exercise
  Interventions: Behavioral: Fasted exercise
- High protein breakfast exercise (Experimental): High protein breakfast consumption prior to exercise
  Interventions: Behavioral: High protein breakfast exercise
- High carbohydrate breakfast exercise (Experimental): High carbohydrate breakfast consumption prior to exercise
  Interventions: Behavioral: High carbohydrate breakfast exercise

INTERVENTIONS:
Behavioral: Fasted exercise — Participants will remain fast (Fasted) 2 h prior to 45 min exercise at 65% VO2max.
  Arms: Fasted exercise
Behavioral: High protein breakfast exercise — Participants will consume a high protein breakfast (Protein) 2 h prior to 45 min exercise at 65% VO2max.
  Arms: High protein breakfast exercise
Behavioral: High carbohydrate breakfast exercise — Participants will consume a high carbohydrate breakfast (Carbohydrate) 2 h prior to 45 min exercise at 65% VO2max.
  Arms: High carbohydrate breakfast exercise

SUMMARY:
This project aims to investigate the impact of acute bout of submaximal exercise under different pre-exercise dietary conditions (fasted state versus high carbohydrate breakfast versus high protein breakfast) on postprandial glycaemic, appetite regulation and energy balance in active healthy women.

DETAILED DESCRIPTION:
Participants will be asked to arrive to the laboratory between 08:00 and 9:00 am after not eating for between 12-14 hours i.e. in a fasted state (water intake is permitted and encouraged). Participants will then be given one of three test drinks (i.e., breakfast): 1) water only; 2) high carbohydrate drink; or 3) high protein (whey protein) drink. Each of these drinks will also contain 500 mL of water and artificial sweetener. 2 h after breakfast, participants will then exercise on a treadmill for 45 min followed by a 2-h oral glucose tolerance test (OGTT) and 30 min ad libitum lunch intake. Blood samples, blood pressures and questionnaire (e.g., appetite and mood) will be collected in a regular pattern throughout the trials. Cognitive functions will be tested at baseline, pre-exercise and 2 h post-exercise. Energy balance will be assessed using food diary and an accelerometer for the rest of the day after leaving the laboratory until midnight.

ELIGIBILITY:
Inclusion Criteria:

* Healthy physical active women (self-reported regular exercise at least 30 min moderate-intensity 3 times per week)
* Aged between 30 to 55 years
* Weight stable for more than 3 months (no change in weight +/- 3%)
* Non-smoker

Exclusion Criteria:

* Personal history of/existing diabetes, cardiovascular disease, metabolic disease or dyslipidaemia
* Taking medications that may influence lipid or carbohydrate metabolism or immune system function
* Men
* Physically inactive

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 12 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Metabolic health | 150 minutes
  Changes in postprandial blood glucose and insulin responses (e.g., area under the curve) post-exercise between trials

SECONDARY OUTCOMES:
Lipid profile | 150 minutes
  Changes in blood triglycerides, cholesterol & NEFA concentrations post-exercise between trials
Gut hormones | 150 minutes
  Changes in gut hormones (e.g., GLP-1, PYY and GIP, etc.) responses post-exercise between trials
Appetite | 30 minutes
  ad libitum lunch energy intake (i.e., kcal) after OGTT between trials
Visual analogue scale (VAS) | 305 minutes
  Changes in VAS from 1-100 mm (e.g., appetite & mood, etc.) between trials
Substrate oxidation | 305 minutes
  Changes in total energy expenditure (i.e., kcal), lipid oxidation (i.e., kcal) and carbohydrate oxidation (i.e., kcal) between trials including pre-exercise, during exercise and post-exercise period.
Inflammation | 305 minutes
  Changes in inflammation biomarkers (e.g., IL-6, IL-10 and IL-1ra, etc.) responses during trials
Blood pressure | 305 minutes
  Changes in blood pressure (e.g., systolic and diastolic blood pressure) during trials
Cognition | 305 minutes
  Changes in cognitive performance (e.g., reaction time in milliseconds and accuracy in percentage) during trials
Energy intake | 600 minutes
  Changes in energy intake (e.g, total calories) using food diary once participants leaving the laboratory until midnight
Physical activity level | 600 minutes
  Changes in physical activity level using an accelerometer to record once participants leaving the laboratory until midnight

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Chih Chen, PhD, Principal Investigator — National Taiwan Normal University
Locations (1):
- National Taiwan Normal University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No